CLINICAL TRIAL: NCT00869284
Title: Phase II Study Treatment of High Risk Non-Hodgkin's Lymphomas
Brief Title: Long-Term Follow-up of Tandem High-Dose Therapy With Peripheral Blood Stem Cell for Adults With High-Risk Age-Adjusted IPI Aggressive Non-Hodgkin's Lymphomas
Acronym: 073
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Amgen (Industry)
Responsible Party: Pr Noel MILPIED, Groupe Ouest Est des Leucémies et autres maladies du sang
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOELAMS 073; no other identification number
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Lymphoma
Keywords: High-dose chemotherapy; aggressive NHL; high-risk; PBSC
MeSH Terms: conditions — Lymphoma | interventions — TANDEM (quinoxaline); Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: CEEP regimen — cyclophosphamide 1200 mg/m² intravenously on day 1 (d1), epirubicin 100 mg/m² intravenously on d1, vindesine 3 mg/m² intravenously on d1 and prednisone 80 mg/m² orally or intravenously on d1-5, with two weeks intervals
Procedure: Tandem high-dose therapy (HDT) followed by autologous peripheral blood stem cell (PBSC) — The conditioning regimen of the first HDT was mitoxantrone 45 mg/m² intravenously on d1 + cytarabine 1000 mg/m² by a 3-hour infusion every 12 hours from d1-4.
  The conditioning regimen of the second HDT started d30 to d45 after the first stem cell infusion, and consisted of 1200 cGy total body irradiation (TBI) in 6 twice daily 200 cGy fractionated doses with a 800 cGy pulmonary shielding, followed by CBV: carmustine 300 mg/m² intravenously on d4, etoposide 200 mg/m² intravenously on d5-8 and cyclophosphamide 1500 mg/m² intravenously on d5-8.

SUMMARY:
Phase II multicenter pilot trial (073) evaluating tandem HDT with PBSC support in aa-IPI=3 untreated aggressive NHL.

DETAILED DESCRIPTION:
High-dose chemotherapy; untreated aggressive non-Hodgkin's lymphoma; high-risk; peripheral blood stem cell support Patients were aged from 15 to 60 years

ELIGIBILITY:
Inclusion Criteria:

* patients aged from 15 to 60 years
* previously untreated
* histologically proven aggressive NHL
* high aa-IPI (equal to 3)
* proper underlying organ function

Exclusion Criteria:

* transformed low-grade, lymphoblastic, mantle-cell, or Burkitt's lymphoma

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 1994-10; Primary Completion 1999-07 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Complete response | end of treatment

SECONDARY OUTCOMES:
overall survival disease free survival | 10 years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Noël MILPIED, MDPD, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Emmanuel Gyan, Tours, France

REFERENCES:
- [Derived] Monjanel H, Deconinck E, Perrodeau E, Gastinne T, Delwail V, Moreau A, Francois S, Berthou C, Gyan E, Milpied N; GOELAMS. Long-term follow-up of tandem high-dose therapy with autologous stem cell support for adults with high-risk age-adjusted international prognostic index aggressive non-Hodgkin Lymphomas: a GOELAMS pilot study. Biol Blood Marrow Transplant. 2011 Jun;17(6):935-40. doi: 10.1016/j.bbmt.2010.11.017. Epub 2010 Nov 23. PMID 21109011